CLINICAL TRIAL: NCT03848845
Title: A Phase I/II Single Arm Open-Label Study to Explore Safety and Clinical Activity of GSK2857916 Administered in Combination With Pembrolizumab in Subjects With Relapsed/Refractory Multiple Myeloma (DREAMM 4)
Brief Title: Study Evaluating Safety, Tolerability and Clinical Activity of GSK2857916 in Combination With Pembrolizumab in Subjects With Relapsed/Refractory Multiple Myeloma (RRMM)
Acronym: DREAMM 4
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 205207; KEYNOTE PN489 (Other: Merck); 2018-002816-29 (EudraCT Number)
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
Keywords: GSK2857916, Pembrolizumab, Multiple Myeloma, RP2D
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Subjects will receive GSK2857916 at escalating doses along with pembrolizumab on Day 1 of each 21-day Cycle to establish RP2D during the Part 1 of the study. Subjects will receive GSK2857916 at RP2D along with pembrolizumab on Day 1 of each 21-day Cycle in Part 2 of the study.
Masking Description: This will be an open-label study. Hence, there will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose escalation (Experimental): Subjects will receive belantamab mafodotin at escalating doses of 2.5 milligrams per kilograms (mg/kg) and 3.4 mg/kg along with 200 mg pembrolizumab via intravenous (IV) infusion on Day 1 of each 21-day cycle to establish RP2D. There will be maximum of 35 cycles of combination treatment.
  Interventions: Drug: belantamab mafodotin; Drug: Pembrolizumab
- Part 2: Expansion cohort (Experimental): Subjects will receive belantamab mafodotin at RP2D along with 200 mg pembrolizumab via IV infusion on Day 1 of each 21-day cycle. There will be maximum of 35 cycles of combination treatment.
  Interventions: Drug: belantamab mafodotin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: belantamab mafodotin — belantamab mafodotin will be available as 20 milligrams per millilitre (mg/mL) solution for IV infusion, supplied as frozen liquid. belantamab mafodotin solution will be diluted in normal 0.9% saline to the appropriate concentration for the dose.
Drug: Pembrolizumab — Pembrolizumab will be available as 100 mg/4 mL solution that should be stored under refrigeration at 2-8 degree Celsius. Pembrolizumab injection (solution) will be diluted prior to IV administration in 0.9% sodium chloride injection or 5% dextrose injection.

SUMMARY:
This is a phase I/II, single arm, open label, two-part study that will assess safety, tolerability and clinical activity of GSK2857916 given in combination with a programmed cell death-1 (PD-1) inhibitor pembrolizumab in subjects with RRMM. This study will enroll adult subjects with RRMM, who have undergone stem cell transplant or who are considered transplant ineligible. Part 1 is a dose escalation phase to evaluate the safety and tolerability of escalating doses of GSK2857916 in combination with 200 milligrams (mg) pembrolizumab to establish the recommended phase 2 dose (RP2D). The following dose levels of GSK2857916 are planned to be studied: 2.5 milligrams per kilograms (mg/kg) (dose level [DL] 1) and 3.4 mg/kg (DL2). Part 2 is a dose expansion cohort. Once the RP2D has been identified, an expansion cohort will open for enrolment to confirm the safety profile and to evaluate the clinical activity of the combination. Up to 40 evaluable subjects will be enrolled in this two-part study (up to 12 in Part 1, and 28 in Part 2).

ELIGIBILITY:
Inclusion criteria:

* Provide signed written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Male or female, 18 years or older (at the time consent is obtained).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subjects must: have histologically or cytologically confirmed diagnosis of Multiple myeloma (MM), as defined by IMWG, 2014 and has undergone stem cell transplant or is considered transplant ineligible, and has been treated with at least 3 prior lines of prior anti-myeloma treatments including an immunomodulatory imide drug (IMiD) (eg. lenalidomide or pomalidomide), a proteasome inhibitor (eg. bortezomib, ixazomib or carfilzomib) and an anti-CD38 antibody alone or in combination. Line of therapy are defined by consensus panel of the International Myeloma Workshop, Has measurable disease defined as one the following: a) Serum M-protein >=0.5 grams per deciliter (g/dL) (>=5 grams per liter [g/L]). b) Urine M-protein ≥200 mg/24h. c) Serum Free light chain (FLC) assay: Involved FLC level ≥10 milligrams per deciliter (mg/dL) (≥100 milligrams per liter [mg/L]) and an abnormal serum free light chain ratio (<0.26 or >1.65).
* Subjects with a history of autologous stem cell transplant are eligible for study participation provided the following eligibility criteria are met: a) transplant was > 100 days prior to study enrolment. b) no active infection(s). c) subject meets the remainder of the eligibility criteria.
* Adequate organ system functions as defined by the laboratory assessments.
* All prior treatment-related toxicities (defined by National Cancer Institute-Common Toxicity Criteria for Adverse Events [NCI-CTCAE], version 4.03, 2010) must be <= Grade 1 at the time of enrolment except for alopecia and Grade 2 neuropathy.
* A female subject is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: is not a woman of childbearing potential (WOCBP) OR is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, during the intervention period and for at least 120 days after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study intervention. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Male subjects are eligible to participate if they agree to the following during the intervention period and for at least 140 days after the last dose of study intervention. Male subjects should refrain from donating sperm, plus, either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR Must agree to use a male condom and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.

Exclusion criteria:

A subject will NOT be eligible for inclusion in this study if any of the following criteria apply:

* Systemic anti-myeloma therapy or an investigational drug <=14 days or five half-lives, whichever is shorter, preceding the first dose of study drug
* Plasmapheresis within 7 days prior to the first dose of study drug
* Prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs
* Has received prior therapy with an anti-PD-1, anti-Programmed cell death Ligand 1 (PD-L1), or anti-Programmed cell death Ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated antigen 4 [CTLA-4], OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher immune related adverse event (irAE)
* Current corneal epithelial disease except mild punctate keratopathy
* Any major surgery within the last four weeks prior to the first dose of study therapy
* Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect subject's safety). Subjects with isolated proteinuria resulting from MM are eligible, provided they fulfil criteria as per adequate organ system function mentioned under inclusion criteria.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Has received prior radiotherapy within 2 weeks of start of study therapy. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (<=2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
* History of (non-infectious) pneumonitis that required steroids, or current pneumonitis
* Current active liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Malignancies other than disease under study are excluded, except for any other malignancy from which the subject has been disease-free for more than 2 years and, in the opinion of the principal investigators and GSK Medical Monitor, will not affect the evaluation of the effects of this clinical trial treatment on the currently targeted malignancy (RRMM). Subjects with curatively treated non-melanoma skin cancer are allowed.
* Has known active CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study therapy
* Evidence of cardiovascular risk including any of the following: a) corrected for heart rate by Fridericia's formula (QTcF) interval ≥470 msecs. b) Evidence of current clinically significant uncontrolled arrhythmias; i. including clinically significant ECG abnormalities including 2nd degree (Type II) or 3rd degree atrioventricular (AV) block. c) History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within six months of Screening. d) Class III or IV heart failure as defined by the New York Heart Association functional classification system. e) Uncontrolled hypertension. f) Presence of cardiac pacemaker (or defibrillator) with a predominantly ventricular paced rhythm, limiting ECG/QTcF analysis. g) Abnormal cardiac valve morphology (>=Grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GSK2857916 or pembrolizumab, or any of the components of the study treatment.
* Pregnant or lactating female.
* Known active infection requiring antibiotic, antiviral, or antifungal treatment.
* Known Human Immunodeficiency Virus (HIV) infection.
* Presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb) at screening or within 3 months prior to first dose of study treatment
* Positive hepatitis C antibody test result or positive hepatitis C Ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* Has received a live-virus vaccination within 30 days of planned start of study therapy.
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other chronic form of immunosuppressive therapy within 7 days prior the first dose of study therapy.
* Has known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (4):
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Madison, Wisconsin
- Canada (2):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Toronto, Ontario
- Germany (3):
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Spain (3):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Suvannasankha A, Bahlis N, Trudel S, Weisel K, Koenecke C, Oriol A, Voorhees PM, Alonso AA, Callander NS, Mateos MV, Reddy N, Hakim S, LaMacchia J, Patel N, Williams D, Jewell RC, Zhou X, Gupta I, Opalinska J, Nooka AK. Safety and efficacy of belantamab mafodotin with pembrolizumab in patients with relapsed or refractory multiple myeloma. Cancer. 2024 Aug 1;130(15):2629-2641. doi: 10.1002/cncr.35319. Epub 2024 Apr 17. PMID 38630908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of two phases - Main Study Phase and Post Analysis Continued Treatment (PACT) Phase. In PACT phase those participants still benefiting from drug continued to receive study drug until discontinued or withdrawn from study.
Pre-assignment Details: Total of 41 participants were enrolled in this study.
Groups:
- Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation: Participants were administered 2.5 mg/kg of belantamab mafodotin in combination with 200 mg of pembrolizumab via intravenous (IV) infusion on Day 1 of each 21-day Cycle up to until disease progression, intolerable toxicity, informed consent withdrawal , or for a maximum of 35 cycles.
- Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation: Participants were administered with 3.4 mg/kg of belantamab mafodotin in combination with 200 mg of pembrolizumab via IV infusion on Day 1 of each 21-day Cycle up to until disease progression, intolerable toxicity, informed consent withdrawal, or for a maximum of 35 cycles.
- Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion: Participants were administered belantamab mafodotin with recommended phase 2 dose (RP2D) of 2.5 mg/kg in combination with 200 mg of pembrolizumab via IV infusion on Day 1 of each 21-day Cycle up to until disease progression, intolerable toxicity, informed consent withdrawal, or for a maximum of 35 cycles.
- PACT Phase- Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg: Participants who completed approximately 178 weeks of treatment of 2.5 mg/kg belantamab mafodotin in combination with 200 mg of pembrolizumab via IV infusion had the opportunity to continue receiving belantamab mafodotin in the PACT phase up to approximately 221 weeks.
Period: Main Study Phase (Day 1 to Week 178)
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion | PACT Phase- Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg
Started | 6 | 7 | 28 | 0
Completed (Participants who completed follow-up or who died were considered to have completed the study.) | 3 (1 participant completed follow-up and 2 participants died) | 4 (1 participant completed follow-up and 3 participants died) | 19 (12 participants completed follow-up and 7 participants died) | 0
Not Completed | 3 | 3 | 9 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 8 | 0
Period: PACT Phase (Week 178 to Week 221)
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion | PACT Phase- Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg
Started | 0 | 0 | 0 | 2
Completed | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion | Total
Number analyzed (Participants) | 6 | 7 | 28 | 41
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 66.8 (12.09) | 67.7 (9.21) | 61.5 (9.41) | 63.3 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 10 | 19
  Male | 1 | 3 | 18 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 1
  Black OR African American | 1 | 2 | 4 | 7
  White | 5 | 5 | 23 | 33

OUTCOME MEASURES:

1. Primary Outcome: Part 1 - Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function.
Time Frame: Up to approximately 31 months
Population: All Treated Population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 6 | 7
Participants
  AEs | 6 | 7
  SAEs | 4 | 5

2. Primary Outcome: Part 1 - Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT is an AE that is considered by the investigator to be clinically relevant and attributed to the study therapy during the 21 day DLT period and meets at least one of the DLT criteria: any Grade 4 and 3 non-hematologic toxicity, any Grade 3 or greater non-hematologic laboratory value, hematologic toxicity lasting >=7 days, except Grade 4 thrombocytopenia of any duration or Grade 3 thrombocytopenia associated with clinically significant bleeding. Grade 3 or greater febrile neutropenia lasting >48 hours (h) despite adequate treatment, Nephrotoxicity requiring dialysis, Liver toxicity, prolonged delay (>14 days) in initiating Cycle 2 due to any treatment (pembrolizumab or GSK2857916) related toxicity, any treatment-related toxicity that causes discontinuation of treatment during Cycle 1, any other toxicity considered to be dose-limiting that occurs beyond 21 days and any other event which in the judgment of the investigator and GlaxoSmithKline Medical Monitor is considered to be a DLT.
Time Frame: Up to 21 days
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 6 | 7
Participants | 0 | 0

3. Primary Outcome: Part 1 - Number of Participants With Worst-case Grade Change From Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: hemoglobin, White blood cells (WBC) count, lymphocytes, neutrophils and platelet count. The laboratory parameters were graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Any worst-case post baseline increase in grade along with any increase to a maximum grade of 3 and a maximum grade of 4 are presented.
Time Frame: Baseline (Day 1) and up to approximately 31 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 6 | 7
Participants
  Hemoglobin Decreased (Anemia), Any Grade Increase | 4 | 2
  Hemoglobin Decreased (Anemia), Increase to Grade 3 | 3 | 1
  Hemoglobin Decreased (Anemia), Increase to Grade 4 | 0 | 0
  Hemoglobin Increased, Any Grade Increase | 0 | 0
  Hemoglobin Increased, Increase to Grade 3 | 0 | 0
  Hemoglobin Increased, Increase to Grade 4 | 0 | 0
  WBC Increased (Leukocytosis), Any Grade Increase | 0 | 0
  WBC Increased (Leukocytosis), Increase to Grade 3 | 0 | 0
  WBC Increased (Leukocytosis), Increase to Grade 4 | 0 | 0
  WBC Decreased, Any Grade Increase | 3 | 3
  WBC Decreased, Increase to Grade 3 | 1 | 1
  WBC Decreased, Increase to Grade 4 | 0 | 0
  Lymphocyte Decreased, Any Grade Increase | 4 | 1
  Lymphocyte Decreased, Increase to Grade 3 | 1 | 1
  Lymphocyte Decreased, Increase to Grade 4 | 1 | 0
  Lymphocyte Increased, Any Grade Increase | 0 | 1
  Lymphocyte Increased, Increase to Grade 3 | 0 | 0
  Lymphocyte Increased, Increase to Grade 4 | 0 | 0
  Neutrophil Decreased, Any Grade Increase | 5 | 2
  Neutrophil Decreased, Increase to Grade 3 | 2 | 1
  Neutrophil Decreased, Increase to Grade 4 | 0 | 1
  Platelet Decreased, Any Grade Increase | 5 | 5
  Platelet Decreased, Increase to Grade 3 | 3 | 3
  Platelet Decreased, Increase to Grade 4 | 1 | 0

4. Primary Outcome: Part 1 - Number of Participants With Worst-case Change Post-baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: basophils, eosinophils, mean corpuscular hemoglobin concentration (MCHC), mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), erythrocytes, hematocrit, monocytes, neutrophils and reticulocyte. The summaries of worst-case change from baseline with respect to normal range was analyzed for only those laboratory tests that were not gradable by CTCAE version 4.03. The number of participants with decreases to low from baseline, changes to normal or no changes from baseline, and increases to high values have been presented.
Time Frame: Baseline (Day 1) and up to approximately 31 months
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 6 | 7
Participants
  Basophils, Decrease to Low: number analyzed (Participants) | 6 | 6
  Basophils, Decrease to Low | 0 | 0
  Basophils, Change to Normal or No Change: number analyzed (Participants) | 6 | 6
  Basophils, Change to Normal or No Change | 6 | 6
  Basophils, Increase to High: number analyzed (Participants) | 6 | 6
  Basophils, Increase to High | 0 | 0
  Eosinophils, Decrease to Low | 2 | 1
  Eosinophils, Change to Normal or No Change | 4 | 6
  Eosinophils, Increase to High | 0 | 0
  MCHC, Decrease to Low | 0 | 1
  MCHC, Change to Normal or No Change | 6 | 4
  MCHC, Increase to High | 0 | 2
  MCH, Decrease to Low: number analyzed (Participants) | 5 | 6
  MCH, Decrease to Low | 2 | 0
  MCH, Change to Normal or No Change: number analyzed (Participants) | 5 | 6
  MCH, Change to Normal or No Change | 3 | 5
  MCH, Increase to High: number analyzed (Participants) | 5 | 6
  MCH, Increase to High | 0 | 1
  MCV, Decrease to Low | 1 | 0
  MCV, Change to Normal or No Change | 5 | 6
  MCV, Increase to High | 0 | 1
  Erythrocytes, Decrease to Low | 0 | 1
  Erythrocytes, Change to Normal or No Change | 6 | 6
  Erythrocytes, Increase to High | 0 | 0
  Hematocrit, Decrease to Low | 0 | 0
  Hematocrit, Change to Normal or No Change | 5 | 7
  Hematocrit, Increase to High | 1 | 0
  Monocytes, Decrease to Low | 0 | 0
  Monocytes, Change to Normal or No Change | 3 | 4
  Monocytes, Increase to High | 3 | 3
  Neutrophils, Decrease to Low: number analyzed (Participants) | 0 | 0
  Neutrophils, Change to Normal or No Change: number analyzed (Participants) | 0 | 0
  Neutrophils, Increase to High: number analyzed (Participants) | 0 | 0
  Reticulocyte, Decrease to Low: number analyzed (Participants) | 6 | 6
  Reticulocyte, Decrease to Low | 4 | 0
  Reticulocyte, Change to Normal or No Change: number analyzed (Participants) | 6 | 6
  Reticulocyte, Change to Normal or No Change | 0 | 4
  Reticulocyte, Increase to High: number analyzed (Participants) | 6 | 6
  Reticulocyte, Increase to High | 4 | 2

5. Primary Outcome: Part 1 - Number of Participants With Worst-case Grade Change From Baseline in Lab Chemistry Parameters
Description: Blood samples were collected for the analysis of clinical chemistry parameters: glucose, alanine aminotransferase (ALT), albumin, alkaline phosphatase, aspartate aminotransferase (AST), blood bilirubin, calcium, creatine kinase (CPK), creatinine, gamma glutamyl transferase (GGT), magnesium, phosphate, potassium and sodium. Laboratory parameters were graded according to NCI-CTCAE version 4.03. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Any worst case post baseline increase in grade along with any increase to a maximum grade of 3 and a maximum grade of 4 are presented.
Time Frame: Baseline (Day 1) and up to approximately 31 months
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 6 | 7
Participants
  Glucose Increased (Hyperglycemia), Any Grade Increase: number analyzed (Participants) | 5 | 5
  Glucose Increased (Hyperglycemia), Any Grade Increase | 0 | 0
  Glucose Increased (Hyperglycemia), Increase to Grade 3: number analyzed (Participants) | 5 | 5
  Glucose Increased (Hyperglycemia), Increase to Grade 3 | 0 | 0
  Glucose Increased (Hyperglycemia), Increase to Grade 4: number analyzed (Participants) | 5 | 5
  Glucose Increased (Hyperglycemia), Increase to Grade 4 | 0 | 0
  Glucose Decreased (Hypoglycemia), Any Grade Increase: number analyzed (Participants) | 5 | 5
  Glucose Decreased (Hypoglycemia), Any Grade Increase | 1 | 0
  Glucose Decreased (Hypoglycemia), Increase to Grade 3: number analyzed (Participants) | 5 | 5
  Glucose Decreased (Hypoglycemia), Increase to Grade 3 | 0 | 0
  Glucose Decreased (Hypoglycemia), Increase to Grade 4: number analyzed (Participants) | 5 | 5
  Glucose Decreased (Hypoglycemia), Increase to Grade 4 | 0 | 0
  ALT Increased, Any Grade Increase | 3 | 0
  ALT Increased, Increase to Grade 3 | 0 | 0
  ALT Increased, Increase to Grade 4 | 0 | 0
  Albumin Decreased (Hypoalbuminemia), Any Grade Increase | 1 | 4
  Albumin Decreased (Hypoalbuminemia), Increase to Grade 3 | 0 | 0
  Albumin Decreased (Hypoalbuminemia), Increase to Grade 4 | 0 | 0
  Alkaline phosphatase Increased, Any Grade Increase | 3 | 2
  Alkaline phosphatase Increased, Increase to Grade 3 | 0 | 0
  Alkaline phosphatase Increased, Increase to Grade 4 | 0 | 0
  AST Increased, Any Grade Increase | 5 | 5
  AST Increased, Increase to Grade 3 | 0 | 0
  AST Increased, Increase to Grade 4 | 0 | 0
  Blood bilirubin Increased, Any Grade Increase | 0 | 1
  Blood bilirubin Increased, Increase to Grade 3 | 0 | 0
  Blood bilirubin Increased, Increase to Grade 4 | 0 | 0
  Calcium Increased (Hypercalcemia), Any Grade Increase: number analyzed (Participants) | 5 | 4
  Calcium Increased (Hypercalcemia), Any Grade Increase | 2 | 1
  Calcium Increased (Hypercalcemia), Increase to Grade 3: number analyzed (Participants) | 5 | 4
  Calcium Increased (Hypercalcemia), Increase to Grade 3 | 0 | 0
  Calcium Increased (Hypercalcemia), Increase to Grade 4: number analyzed (Participants) | 5 | 4
  Calcium Increased (Hypercalcemia), Increase to Grade 4 | 0 | 0
  Calcium Decreased (Hypocalcemia), Any Grade Increase: number analyzed (Participants) | 5 | 4
  Calcium Decreased (Hypocalcemia), Any Grade Increase | 2 | 0
  Calcium Decreased (Hypocalcemia), Increase to Grade 3: number analyzed (Participants) | 5 | 4
  Calcium Decreased (Hypocalcemia), Increase to Grade 3 | 0 | 0
  Calcium Decreased (Hypocalcemia), Increase to Grade 4: number analyzed (Participants) | 5 | 4
  Calcium Decreased (Hypocalcemia), Increase to Grade 4 | 0 | 0
  CPK Increased, Any Grade Increase | 1 | 2
  CPK Increased, Increase to Grade 3 | 0 | 0
  CPK Increased, Increase to Grade 4 | 0 | 0
  Creatinine Increased, Any Grade Increase | 2 | 1
  Creatinine Increased, Increase to Grade 3 | 0 | 0
  Creatinine Increased, Increase to Grade 4 | 0 | 0
  GGT Increased, Any Grade Increase | 3 | 2
  GGT Increased, Increase to Grade 3 | 0 | 0
  GGT Increased, Increase to Grade 4 | 0 | 0
  Magnesium Increased (Hypermagnesemia), Any Grade Increase | 0 | 0
  Magnesium Increased (Hypermagnesemia), Increase to Grade 3 | 0 | 0
  Magnesium Increased (Hypermagnesemia), Increase to Grade 4 | 0 | 0
  Magnesium Decreased (Hypomagnesemia), Any Grade Increase | 2 | 2
  Magnesium Decreased (Hypomagnesemia), Increase to Grade 3 | 0 | 0
  Magnesium Decreased (Hypomagnesemia), Increase to Grade 4 | 0 | 0
  Phosphate Decreased (Hypophosphatemia), Any Grade Increase | 2 | 0
  Phosphate Decreased (Hypophosphatemia), Increase to Grade 3 | 0 | 0
  Phosphate Decreased (Hypophosphatemia), Increase to Grade 4 | 0 | 0
  Potassium Increased (Hyperkalemia), Any Grade Increase | 0 | 0
  Potassium Increased (Hyperkalemia), Increase to Grade 3 | 0 | 0
  Potassium Increased (Hyperkalemia), Increase to Grade 4 | 0 | 0
  Potassium Decreased (Hypokalemia), Any Grade Increase | 2 | 2
  Potassium Decreased (Hypokalemia), Increase to Grade 3 | 0 | 1
  Potassium Decreased (Hypokalemia), Increase to Grade 4 | 0 | 0
  Sodium Increased (Hypernatremia), Any Grade Increase | 0 | 0
  Sodium Increased (Hypernatremia), Increase to Grade 3 | 0 | 0
  Sodium Increased (Hypernatremia), Increase to Grade 4 | 0 | 0
  Sodium Decreased (Hyponatremia), Any Grade Increase | 1 | 3
  Sodium Decreased (Hyponatremia), Increase to Grade 3 | 0 | 2
  Sodium Decreased (Hyponatremia), Increase to Grade 4 | 0 | 0

6. Primary Outcome: Part 1 - Number of Participants With Worst-case Change Post-baseline in Lab Chemistry Parameters
Description: Blood samples were collected for the analysis of following chemistry parameters: calcium, carbon dioxide, chloride, direct bilirubin, protein, thyrotropin (TSH), thyroxine (T4) and triiodothyronine (T3). The summaries of worst case change from baseline with respect to normal range was analyzed for only those laboratory tests that were not gradable by CTCAE version 4.03. The number of participants with decreases to low from baseline, changes to normal or no changes from baseline, and increases to high values have been presented.
Time Frame: Baseline (Day 1) and up to 31 months
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 6 | 7
Participants
  Calcium, Decrease to Low | 1 | 2
  Calcium, Change to Normal or No Change | 4 | 4
  Calcium, Increase to High | 1 | 1
  Carbon dioxide, Decrease to Low: number analyzed (Participants) | 6 | 6
  Carbon dioxide, Decrease to Low | 2 | 1
  Carbon dioxide, Change to Normal or No Change: number analyzed (Participants) | 6 | 6
  Carbon dioxide, Change to Normal or No Change | 3 | 4
  Carbon dioxide, Increase to High: number analyzed (Participants) | 6 | 6
  Carbon dioxide, Increase to High | 1 | 1
  Chloride, Decrease to Low | 1 | 2
  Chloride, Change to Normal or No Change | 4 | 4
  Chloride, Increase to High | 1 | 1
  Direct bilirubin, Decrease to Low: number analyzed (Participants) | 5 | 6
  Direct bilirubin, Decrease to Low | 0 | 0
  Direct bilirubin, Change to Normal or No Change: number analyzed (Participants) | 5 | 6
  Direct bilirubin, Change to Normal or No Change | 4 | 5
  Direct bilirubin, Increase to High: number analyzed (Participants) | 5 | 6
  Direct bilirubin, Increase to High | 1 | 1
  Protein, Decrease to Low | 2 | 3
  Protein, Change to Normal or No Change | 3 | 4
  Protein, Increase to High | 1 | 1
  TSH, Decrease to Low: number analyzed (Participants) | 6 | 6
  TSH, Decrease to Low | 0 | 0
  TSH, Change to Normal or No Change: number analyzed (Participants) | 6 | 6
  TSH, Change to Normal or No Change | 3 | 4
  TSH, Increase to High: number analyzed (Participants) | 6 | 6
  TSH, Increase to High | 3 | 2
  T4, Decrease to Low: number analyzed (Participants) | 6 | 6
  T4, Decrease to Low | 1 | 0
  T4, Change to Normal or No Change: number analyzed (Participants) | 6 | 6
  T4, Change to Normal or No Change | 5 | 6
  T4, Increase to High: number analyzed (Participants) | 6 | 6
  T4, Increase to High | 1 | 0
  T3, Decrease to Low: number analyzed (Participants) | 2 | 1
  T3, Decrease to Low | 1 | 1
  T3, Change to Normal or No Change: number analyzed (Participants) | 2 | 1
  T3, Change to Normal or No Change | 1 | 0
  T3, Increase to High: number analyzed (Participants) | 2 | 1
  T3, Increase to High | 0 | 0

7. Primary Outcome: Part 1 - Number of Participants With Worst-case Change Post-baseline Urinalysis Results
Description: Urine samples were collected to assess urine glucose, protein, occult blood and ketones using dipstick method. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as negative, trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Result for urinalysis parameters were recorded as no change/decreased and any increase. Data for worst-case post baseline urinalysis results is presented.
Time Frame: Baseline (Day 1) and up to approximately 31 months
Population: All Treated Population. Only those participants with data available for worst-case post baseline have been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 6 | 7
Participants
  Glucose, No Change/Decreased: number analyzed (Participants) | 6 | 6
  Glucose, No Change/Decreased | 6 | 5
  Glucose, Any Increase: number analyzed (Participants) | 6 | 6
  Glucose, Any Increase | 0 | 1
  Ketones, No Change/Decreased: number analyzed (Participants) | 6 | 6
  Ketones, No Change/Decreased | 3 | 5
  Ketones, Any Increase: number analyzed (Participants) | 6 | 6
  Ketones, Any Increase | 3 | 1
  Occult Blood, No Change/Decreased: number analyzed (Participants) | 6 | 5
  Occult Blood, No Change/Decreased | 4 | 4
  Occult Blood, Any Increase: number analyzed (Participants) | 6 | 5
  Occult Blood, Any Increase | 2 | 1
  Protein, No Change/Decreased: number analyzed (Participants) | 6 | 6
  Protein, No Change/Decreased | 4 | 4
  Protein, Any Increase: number analyzed (Participants) | 6 | 6
  Protein, Any Increase | 2 | 2

8. Primary Outcome: Part 1 - Changes From Baseline in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected from participants to assess urine pH levels. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Baseline (Day 1) and Week 46
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Potential of Hydrogen (pH)
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 2 | 1
Potential of Hydrogen (pH) | 1.0 (2.83) | 0.0

9. Primary Outcome: Part 1 - Changes From Baseline in Urine Specific Gravity
Description: Urine samples were collected from participants to assess urine specific gravity. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Baseline (Day 1) and Week 46
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 2 | 1
Ratio | -0.0010 (0.00566) | 0.0100

10. Primary Outcome: Part 1 - Number of Participants With Worst-case Grade Change From Baseline in Vital Signs: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: DBP and SBP were measured after resting for at least 5 minutes in a supine or semi-recumbent position. They were graded according to NCI-CTCAE version 4.03. For SBP: Grade 0 (<=120 millimeter of mercury [mmHg]), Grade 1 (121-139 mmHg), Grade 2 (140-159 mmHg), Grade 3 (>=160 mmHg). For DBP: Grade 0 (<=80 mmHg), Grade 1 (81-89 mmHg), Grade 2 (90-99 mmHg), Grade 3 (>=100 mmHg). Higher grade indicates greater severity. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst-case post baseline with any grade increase and a maximum post-baseline grade increase to Grade 3 from their baseline grade are presented.
Time Frame: Baseline (Day 1) and up to approximately 31 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 6 | 7
Participants
  DBP, Any Grade Increase | 6 | 4
  DBP, Increase to Grade 2 | 2 | 1
  DBP, Increase to Grade 3 | 0 | 0
  SBP, Any Grade Increase | 6 | 5
  SBP, Increase to Grade 2 | 3 | 2
  SBP, Increase to Grade 3 | 0 | 3

11. Primary Outcome: Part 1 - Number of Participants With Worst-case Change From Baseline in Vital Signs: Pulse Rate and Body Temperature
Description: Vital signs (pulse rate and temperature) were measured after resting for at least 5 minutes in a supine or semi-recumbent position. The abnormal vital sign ranges were: For pulse rate (low <60 beats per minute [bpm] and high >100 bpm); For body temperature (<=35 degrees Celsius or >=38 degrees Celsius). Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst case change from baseline was presented as Baseline to low, Baseline to Normal or No change and Baseline to High.
Time Frame: Baseline (Day 1) and up to approximately 31 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 6 | 7
Participants
  Pulse Rate: Baseline To Low | 3 | 2
  Pulse Rate: Baseline To Normal or No Change | 3 | 3
  Pulse Rate: Baseline To High | 0 | 2
  Temperature: Baseline To Low | 0 | 1
  Temperature: Baseline To Normal or No Change | 4 | 6
  Temperature: Baseline To High | 2 | 0

12. Primary Outcome: Part 2 - Percentage of Participants With Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed partial response (PR) or better (i.e., PR, very good partial response [VGPR], complete response [CR] and stringent complete response [sCR]), according to the International Myeloma Working Group (IMWG) Response Criteria. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=stringent complete response, CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 h.
Time Frame: Up to approximately 31 months
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Percentage of Participants | 43 [24.5 to 62.8]

13. Secondary Outcome: Part 1 - Percentage of Participants With Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed PR or better (i.e., PR, VGPR, CR and sCR), according to the IMWG Response Criteria. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=stringent complete response, CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR >= 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR = >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 h.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation: Participants were administered 3.4 mg/kg of belantamab mafodotin in combination with 200 mg of pembrolizumab via intravenous (IV) infusion on Day 1 of each 21-day Cycle up to until disease progression, intolerable toxicity, informed consent withdrawal , or for a maximum of 35 cycles.
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 6 | 7
Percentage of Participants | 67 [22.3 to 95.7] | 43 [9.9 to 81.6]

14. Secondary Outcome: Part 2 - Number of Participants With AEs and SAEs
Description: as for outcome 1
Time Frame: Up to approximately 178 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Participants
  AEs | 27
  SAEs | 5

15. Secondary Outcome: Part 2 - Number of Participants With Worst-case Grade Change From Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: hemoglobin, White blood cell (WBC) count, lymphocytes, neutrophils and platelet. The laboratory parameters were graded according to NCI-CTCAE version 4.03. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Any worst case post baseline increase in grade along with any increase to a maximum grade of 3 and a maximum grade of 4 are presented.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 27
Participants
  Anemia, Any Grade Increase | 10
  Anemia, Increase to Grade 3 | 3
  Anemia, Increase to Grade 4 | 0
  Hemoglobin increased, Any Grade Increase | 2
  Hemoglobin increased, Increase to Grade 3 | 0
  Hemoglobin increased, Increase to Grade 4 | 0
  Leukocytosis, Any Grade Increase | 1
  Leukocytosis, Increase to Grade 3 | 0
  Leukocytosis, Increase to Grade 4 | 0
  WBC decreased, Any Grade Increase | 11
  WBC decreased, Increase to Grade 3 | 1
  WBC decreased, Increase to Grade 4 | 2
  Lymphocyte count decreased, Any Grade Increase | 14
  Lymphocyte count decreased, Increase to Grade 3 | 3
  Lymphocyte count decreased, Increase to Grade 4 | 4
  Lymphocyte count increased, Any Grade Increase | 2
  Lymphocyte count increased, Increase to Grade 3 | 1
  Lymphocyte count increased, Increase to Grade 4 | 0
  Neutrophil count decreased, Any Grade Increase | 9
  Neutrophil count decreased, Increase to Grade 3 | 1
  Neutrophil count decreased, Increase to Grade 4 | 2
  Platelet count decreased, Any Grade Increase | 18
  Platelet count decreased, Increase to Grade 3 | 7
  Platelet count decreased, Increase to Grade 4 | 4

16. Secondary Outcome: Part 2 - Number of Participants With Worst-case Change Post-baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: basophils, eosinophils, mean corpuscular hemoglobin concentration (MCHC), mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), Erythrocytes, hematocrit, monocytes, neutrophils and reticulocyte. The summaries of worst-case change from baseline with respect to normal range was analyzed for only those laboratory tests that were not gradable by CTCAE version 4.03. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. The number of participants with decreases to low from baseline, changes to normal or no changes from baseline, and increases to high values have been presented.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 27
Participants
  Basophils, Decrease to Low: number analyzed (Participants) | 23
  Basophils, Decrease to Low | 0
  Basophils, Change to Normal or No Change: number analyzed (Participants) | 23
  Basophils, Change to Normal or No Change | 22
  Basophils, Increase to High: number analyzed (Participants) | 23
  Basophils, Increase to High | 1
  Eosinophils, Decrease to Low: number analyzed (Participants) | 26
  Eosinophils, Decrease to Low | 2
  Eosinophils, Change to Normal or No Change: number analyzed (Participants) | 26
  Eosinophils, Change to Normal or No Change | 22
  Eosinophils, Increase to High: number analyzed (Participants) | 26
  Eosinophils, Increase to High | 3
  MCHC, Decrease to Low | 3
  MCHC, Change to Normal or No Change | 24
  MCHC, Increase to High | 0
  MCH, Decrease to Low: number analyzed (Participants) | 22
  MCH, Decrease to Low | 3
  MCH, Change to Normal or No Change: number analyzed (Participants) | 22
  MCH, Change to Normal or No Change | 16
  MCH, Increase to High: number analyzed (Participants) | 22
  MCH, Increase to High | 3
  MCV, Decrease to Low | 0
  MCV, Change to Normal or No Change | 25
  MCV, Increase to High | 2
  Erythrocytes, Decrease to Low | 0
  Erythrocytes, Change to Normal or No Change | 26
  Erythrocytes, Increase to High | 1
  Hematocrit, Decrease to Low | 3
  Hematocrit, Change to Normal or No Change | 23
  Hematocrit, Increase to High | 1
  Monocytes, Decrease to Low | 0
  Monocytes, Change to Normal or No Change | 20
  Monocytes, Increase to High | 7
  Neutrophils, Segmented, Decrease to Low: number analyzed (Participants) | 1
  Neutrophils, Segmented, Decrease to Low | 0
  Neutrophils, Segmented, Change to Normal or No Change: number analyzed (Participants) | 1
  Neutrophils, Segmented, Change to Normal or No Change | 1
  Neutrophils, Segmented, Increase to High: number analyzed (Participants) | 1
  Neutrophils, Segmented, Increase to High | 0
  Reticulocytes, Decrease to Low: number analyzed (Participants) | 21
  Reticulocytes, Decrease to Low | 2
  Reticulocytes, Change to Normal or No Change: number analyzed (Participants) | 21
  Reticulocytes, Change to Normal or No Change | 14
  Reticulocytes, Increase to High: number analyzed (Participants) | 21
  Reticulocytes, Increase to High | 5

17. Secondary Outcome: Part 2 - Number of Participants With Worst-case Grade Change From Baseline in Lab Chemistry Parameters
Description: Blood samples were collected for the analysis of clinical chemistry parameters: glucose, alanine aminotransferase (ALT), albumin, alkaline phosphatase, aspartate aminotransferase (AST), blood bilirubin, calcium, creatine kinase (CPK), creatinine, gamma glutamyl transferase (GGT), magnesium, phosphate potassium and sodium. Laboratory parameters were graded according to NCI-CTCAE version 4.03. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Higher grade indicates greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Any worst case post baseline increase in grade along with any increase to a maximum grade of 3 and a maximum grade of 4 are presented.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 27
Participants
  Hyperglycemia, Any Grade Increase: number analyzed (Participants) | 23
  Hyperglycemia, Any Grade Increase | 1
  Hyperglycemia, Increase to Grade 3: number analyzed (Participants) | 23
  Hyperglycemia, Increase to Grade 3 | 0
  Hyperglycemia, Increase to Grade 4: number analyzed (Participants) | 23
  Hyperglycemia, Increase to Grade 4 | 0
  Hypoglycemia, Any Grade Increase: number analyzed (Participants) | 23
  Hypoglycemia, Any Grade Increase | 4
  Hypoglycemia, Increase to Grade 3: number analyzed (Participants) | 23
  Hypoglycemia, Increase to Grade 3 | 0
  Hypoglycemia, Increase to Grade 4: number analyzed (Participants) | 23
  Hypoglycemia, Increase to Grade 4 | 0
  ALT increased, Any Grade Increase | 5
  ALT increased, Increase to Grade 3 | 1
  ALT increased, Increase to Grade 4 | 0
  Hypoalbuminemia, Any Grade Increase | 9
  Hypoalbuminemia, Increase to Grade 3 | 1
  Hypoalbuminemia, Increase to Grade 4 | 0
  Alkaline phosphatase increased, Any Grade Increase | 9
  Alkaline phosphatase increased, Increase to Grade 3 | 1
  Alkaline phosphatase increased, Increase to Grade 4 | 0
  AST increased, Any Grade Increase | 20
  AST increased, Increase to Grade 3 | 1
  AST increased, Increase to Grade 4 | 0
  Blood bilirubin increased, Any Grade Increase | 3
  Blood bilirubin increased, Increase to Grade 3 | 1
  Blood bilirubin increased, Increase to Grade 4 | 0
  Hypercalcemia, Any Grade Increase: number analyzed (Participants) | 17
  Hypercalcemia, Any Grade Increase | 3
  Hypercalcemia, Increase to Grade 3: number analyzed (Participants) | 17
  Hypercalcemia, Increase to Grade 3 | 0
  Hypercalcemia, Increase to Grade 4: number analyzed (Participants) | 17
  Hypercalcemia, Increase to Grade 4 | 0
  Hypocalcemia, Any Grade Increase: number analyzed (Participants) | 17
  Hypocalcemia, Any Grade Increase | 3
  Hypocalcemia, Increase to Grade 3: number analyzed (Participants) | 17
  Hypocalcemia, Increase to Grade 3 | 0
  Hypocalcemia, Increase to Grade 4: number analyzed (Participants) | 17
  Hypocalcemia, Increase to Grade 4 | 0
  CPK increased, Any Grade Increase: number analyzed (Participants) | 26
  CPK increased, Any Grade Increase | 4
  CPK increased, Increase to Grade 3: number analyzed (Participants) | 26
  CPK increased, Increase to Grade 3 | 1
  CPK increased, Increase to Grade 4: number analyzed (Participants) | 26
  CPK increased, Increase to Grade 4 | 0
  Creatinine increased, Any Grade Increase | 7
  Creatinine increased, Increase to Grade 3 | 0
  Creatinine increased, Increase to Grade 4 | 0
  GGT increased, Any Grade Increase | 10
  GGT increased, Increase to Grade 3 | 1
  GGT increased, Increase to Grade 4 | 0
  Hypermagnesemia, Any Grade Increase | 0
  Hypermagnesemia, Increase to Grade 3 | 0
  Hypermagnesemia, Increase to Grade 4 | 0
  Hypomagnesemia, Any Grade Increase | 6
  Hypomagnesemia, Increase to Grade 3 | 0
  Hypomagnesemia, Increase to Grade 4 | 0
  Hypophosphatemia, Any Grade Increase | 3
  Hypophosphatemia, Increase to Grade 3 | 1
  Hypophosphatemia, Increase to Grade 4 | 0
  Hyperkalemia, Any Grade Increase | 0
  Hyperkalemia, Increase to Grade 3 | 0
  Hyperkalemia, Increase to Grade 4 | 0
  Hypokalemia, Any Grade Increase | 4
  Hypokalemia, Increase to Grade 3 | 1
  Hypokalemia, Increase to Grade 4 | 0
  Hypernatremia, Any Grade Increase | 0
  Hypernatremia, Increase to Grade 3 | 0
  Hypernatremia, Increase to Grade 4 | 0
  Hyponatremia, Any Grade Increase | 3
  Hyponatremia, Increase to Grade 3 | 1
  Hyponatremia, Increase to Grade 4 | 0

18. Secondary Outcome: Part 2 - Number of Participants With Worst-case Change Post-baseline in Lab Chemistry Parameters
Description: Blood samples were collected for the analysis of following chemistry parameters: calcium, carbon dioxide, chloride, direct bilirubin, protein, thyrotropin (TSH), thyroxine (T4) and triiodothyronine (T3). Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. The summaries of worst case change from baseline with respect to normal range was analyzed for only those laboratory tests that were not gradable by CTCAE version 4.03. The number of participants with decreases to low, changes to normal or no changes from baseline, and increases to high values have been presented.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed. Participants are counted twice if the participant has values that changed "Decreased to Low" and "Increased to High", so the sum of the percentages may not add to 100% for each row
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 27
Participants
  Calcium, Decrease to Low | 4
  Calcium, Change to Normal or No Change | 18
  Calcium, Increase to High | 5
  Carbon Dioxide, Decrease to Low | 4
  Carbon Dioxide, Change to Normal or No Change | 14
  Carbon Dioxide, Increase to High | 9
  Chloride, Decrease to Low | 4
  Chloride, Change to Normal or No Change | 20
  Chloride, Increase to High | 3
  Direct Bilirubin, Decrease to Low: number analyzed (Participants) | 23
  Direct Bilirubin, Decrease to Low | 2
  Direct Bilirubin, Change to Normal or No Change: number analyzed (Participants) | 23
  Direct Bilirubin, Change to Normal or No Change | 15
  Direct Bilirubin, Increase to High: number analyzed (Participants) | 23
  Direct Bilirubin, Increase to High | 7
  Protein, Decrease to Low | 8
  Protein, Change to Normal or No Change | 18
  Protein, Increase to High | 2
  TSH, Decrease to Low: number analyzed (Participants) | 26
  TSH, Decrease to Low | 1
  TSH, Change to Normal or No Change: number analyzed (Participants) | 26
  TSH, Change to Normal or No Change | 17
  TSH, Increase to High: number analyzed (Participants) | 26
  TSH, Increase to High | 8
  T4, Free, Decrease to Low: number analyzed (Participants) | 26
  T4, Free, Decrease to Low | 2
  T4, Free, Change to Normal or No Change: number analyzed (Participants) | 26
  T4, Free, Change to Normal or No Change | 23
  T4, Free, Increase to High: number analyzed (Participants) | 26
  T4, Free, Increase to High | 1
  T3, Decrease to Low: number analyzed (Participants) | 0
  T3, Change to Normal or No Change: number analyzed (Participants) | 0
  T3, Increase to High: number analyzed (Participants) | 0

19. Secondary Outcome: Part 2 - Number of Participants With Worst-case Change Post-baseline Urinalysis Results
Description: Urine samples were collected to assess urine glucose, protein, occult blood and ketones using dipstick method. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as negative, trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Result for uranalysis parameters were recorded as no change/decreased and any increase. Data for worst-case post baseline are presented.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 26
Participants
  Glucose, No Change/Decreased | 25
  Glucose, Any Increase | 1
  Ketones, No Change/Decreased | 21
  Ketones, Any Increase | 5
  Occult Blood, No Change/Decreased: number analyzed (Participants) | 24
  Occult Blood, No Change/Decreased | 15
  Occult Blood, Any Increase: number analyzed (Participants) | 24
  Occult Blood, Any Increase | 9
  Protein, No Change/Decreased | 20
  Protein, Any Increase | 6

20. Secondary Outcome: Part 2 - Changes From Baseline in Urine Specific Gravity
Description: as for outcome 9
Time Frame: Baseline (Day 1) and until end of treatment (up to 178 weeks)
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 25
Ratio
  Baseline | 1.0171 (0.00965)
  End of Treatment: number analyzed (Participants) | 13
  End of Treatment | -0.0001 (0.00813)

21. Secondary Outcome: Part 2 - Changes From Baseline in Urine pH
Description: as for outcome 8
Time Frame: Baseline (Day 1) and until end of treatment (up to 178 weeks)
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Potential of Hydrogen (pH)
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Potential of Hydrogen (pH)
  Baseline | 5.71 (0.844)
  End of Treatment: number analyzed (Participants) | 15
  End of Treatment | 0.10 (0.687)

22. Secondary Outcome: Part 2 - Number of Participants With Worst-case Grade Change From Baseline in Vital Signs: DBP and SBP
Description: DBP and SBP were measured after resting for at least 5 minutes in a supine or semi-recumbent position. They were graded according to NCI-CTCAE version 4.0. For SBP: Grade 0 (<=120 millimeter of mercury [mmHg]), Grade 1 (121-139 mmHg), Grade 2 (140-159 mmHg), Grade 3 (>=160 mmHg). For DBP: Grade 0 (<=80 mmHg), Grade 1 (81-89 mmHg), Grade 2 (90-99 mmHg), Grade 3 (>=100 mmHg). Higher grade indicates greater severity. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. An increase is defined as an increase in grade relative to Baseline grade. Data for worst-case post Baseline with any grade increase and a maximum post-baseline grade increase to Grade 3 from their baseline grade are presented.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Participants
  DBP, Any Grade Increase | 20
  DBP, Increase to Grade 2 | 12
  DBP, Increase to Grade 3 | 2
  SBP, Any Grade Increase | 24
  SBP, Increase to Grade 2 | 16
  SBP, Increase to Grade 3 | 6

23. Secondary Outcome: Part 2 - Number of Participants With Worst-case Change From Baseline in Vital Signs: Pulse Rate and Body Temperature
Description: Vital signs (pulse rate and temperature) were measured after resting for at least 5 minutes in a supine or semi-recumbent position. The abnormal vital sign ranges were: For pulse rate (low <60 beats per minute [bpm] and high >100 bpm); For body temperature (<=35 degrees Celsius or >=38 degrees Celsius). Participants were counted in the worst case category that their value changed to (low, normal or high), unless there was no change in their category. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Participants
  Pulse Rate, To Low | 10
  Pulse Rate, To Normal or No Change | 11
  Pulse Rate, To High | 7
  Temperature, To Low | 2
  Temperature, To Normal or No Change | 23
  Temperature, To High | 3

24. Secondary Outcome: Part 2 - Number of Participants With Maximum Worst-case Change From Baseline in Best Corrected Visual Acuity Test (BCVA) Scores
Description: BCVA score was calculated based on the Logarithm of the Minimum Angle of Resolution (logMAR score). Any maximum worst-case change from baseline categories are presented for right and left eyes. No change/improved vision is defined as a change from baseline <0.12; a possible worsened vision is defined as a change from baseline >=0.12 to <0.3; a definite worsened vision is defined as a change from baseline >=0.3 logMAR score. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 27
Participants
  Left Eye, No change/improved vision | 14
  Left Eye, Possible worsened vision | 5
  Left Eye, Definite worsened vision | 8
  Right Eye, No change/improved vision | 16
  Right Eye, Possible worsened vision | 4
  Right Eye, Definite worsened vision | 7

25. Secondary Outcome: Part 2 - Time Taken for the Onset of First Occurrence of Worsening in BCVA Score
Description: The time for the onset of any visual acuity event (change from baseline logMAR score >= 0.3 in either eye) was calculated.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 10
Days | 78.0 [37 to 273]

26. Secondary Outcome: Part 2 - Outcome of First Occurrence of Worsening Eye in BCVA Score
Description: The onset of any visual acuity event (change from baseline in logMAR score >= 0.3 in either eye) was considered resolved if the change from baseline in logMAR score was less than 0.3 in both eyes. Participants with resolved and not resolved outcome of the worsening eye were presented.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 10
Participants
  Resolved prior to end of treatment exposure | 7
  Resolved post end of treatment exposure | 2
  Not resolved | 1

27. Secondary Outcome: Part 2 - Duration of First Occurrence of Worsening in BCVA Score
Description: The time from onset of any visual acuity event (change from baseline logMAR score >= 0.3 in either eye) until the event is resolved (change from baseline logMAR score < 0.3 in both eyes) was used to calculate the duration of first occurrence.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 9
Days | 47.0 [3 to 65]

28. Secondary Outcome: Part 2 - Number of Participants According to the Number of Definite Events of Worsening of Vision
Description: A definite worsened vision was defined as a change from baseline >=0.3 logMAR score.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 10
Participants
  One | 6
  Two | 1
  Three or more | 3

29. Secondary Outcome: Part 2 - Number of Participants With Resolution of Post Treatment Exposure Worsening in BCVA Score
Description: The event was considered resolved if the change from baseline in logMAR score < 0.3 in both eyes.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 4
Participants
  Resolved | 2
  Not resolved, follow-up ongoing | 0
  Not resolved, follow-up ended | 2

30. Secondary Outcome: Part 2 - Duration of Resolution Post-treatment Exposure of Worsening in BCVA Score
Description: The time taken for the resolution of worsening eye post treatment exposure. Duration was defined as the time from onset of any visual acuity event (change from baseline logMAR score >= 0.3 in either eye) until the event was considered resolved (change from baseline logMAR score < 0.3 in both eyes). It required at least a one day gap between the resolution of all events from first occurrence to the onset of second occurrence. The end of treatment exposure was defined as 20 days from last infusion date.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 2
Days | 34.5 [22 to 47]

31. Secondary Outcome: Part 2 - Number of Participants With Post-baseline Decline in BCVA to Light Perception or no Light Perception
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population. Data was not collected
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 0

32. Secondary Outcome: Part 2 - Number of Participants With Worst-case Shift From Baseline in Ophthalmological Epithelium Exam
Description: Participants with worst-case shift from baseline in corneal epithelium defects by right eye, left eye and worse eye are presented as normal (N), abnormal (AN) and missing. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Participants
  Right Eye: Baseline N, Post-Baseline N | 3
  Right Eye: Baseline N, Post-Baseline AN | 16
  Right Eye: Baseline AN, Post-Baseline N | 0
  Right Eye: Baseline AN, Post-Baseline AN | 8
  Right Eye: Baseline N, Post-Baseline Missing | 0
  Right Eye: Baseline AN, Post-Baseline Missing | 1
  Left Eye: Baseline N, Post-Baseline N | 2
  Left Eye: Baseline N, Post-Baseline AN | 16
  Left Eye: Baseline AN, Post-Baseline N | 1
  Left Eye: Baseline AN, Post-Baseline AN | 8
  Left Eye: Baseline N, Post-Baseline Missing | 1
  Left Eye: Baseline AN, Post-Baseline Missing | 0
  Worse Eye: Baseline N, Post-Baseline N | 3
  Worse Eye: Baseline N, Post-Baseline AN | 17
  Worse Eye: Baseline AN, Post-Baseline N | 0
  Worse Eye: Baseline AN, Post-Baseline AN | 7
  Worse Eye: Baseline N, Post-Baseline Missing | 1
  Worse Eye: Baseline AN, Post-Baseline Missing | 0

33. Secondary Outcome: Part 2 - Number of Participants With Worst-case Shift From Baseline in Corneal Examinations
Description: Participants with worst-case shift from baseline in corneal examination: corneal ulcer, epithelial microcystic edema, subepithelial haze, corneal neovascularization and microcysts without edema, by right eye (R), left eye (L) and worse eye (W) are presented as yes (Y), no (N) and missing (M). Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Participants
  Corneal ulcer indicator left eye: Baseline N, Post-Baseline N | 23
  Corneal ulcer indicator left eye: Baseline N, Post-Baseline Y | 0
  Corneal ulcer indicator left eye: Baseline N, Post-Baseline Missing | 1
  Corneal ulcer indicator left eye: Baseline Y, Post-Baseline N | 0
  Corneal ulcer indicator left eye: Baseline Y, Post-Baseline Y | 0
  Corneal ulcer indicator left eye: Baseline Y, Post-Baseline Missing | 0
  Corneal ulcer indicator left eye: Baseline Missing, Post-Baseline N | 3
  Corneal ulcer indicator left eye: Baseline Missing, Post-Baseline Y | 0
  Corneal ulcer indicator left eye: Baseline Missing, Post-Baseline Missing | 1
  Corneal ulcer indicator right eye: Baseline N, Post-Baseline N | 21
  Corneal ulcer indicator right eye: Baseline N, Post-Baseline Y | 0
  Corneal ulcer indicator right eye: Baseline N, Post-Baseline Missing | 1
  Corneal ulcer indicator right eye: Baseline Y, Post-Baseline N | 0
  Corneal ulcer indicator right eye: Baseline Y, Post-Baseline Y | 0
  Corneal ulcer indicator right eye: Baseline Y, Post-Baseline Missing | 0
  Corneal ulcer indicator right eye: Baseline Missing, Post-Baseline N | 5
  Corneal ulcer indicator right eye: Baseline Missing, Post-Baseline Y | 0
  Corneal ulcer indicator right eye: Baseline Missing, Post-Baseline Missing | 1
  Corneal ulcer indicator worst eye: Baseline N, Post-Baseline N | 23
  Corneal ulcer indicator worst eye: Baseline N, Post-Baseline Y | 0
  Corneal ulcer indicator worst eye: Baseline N, Post-Baseline Missing | 1
  Corneal ulcer indicator worst eye: Baseline Y, Post-Baseline N | 0
  Corneal ulcer indicator worst eye: Baseline Y, Post-Baseline Y | 0
  Corneal ulcer indicator worst eye: Baseline Y, Post-Baseline Missing | 0
  Corneal ulcer indicator worst eye: Baseline Missing, Post-Baseline N | 3
  Corneal ulcer indicator worst eye: Baseline Missing, Post-Baseline Y | 0
  Corneal ulcer indicator worst eye: Baseline Missing, Post-Baseline Missing | 1
  Epithelial microcystic edema indicator left eye: Baseline N, Post-Baseline N | 17
  Epithelial microcystic edema indicator left eye: Baseline N, Post-Baseline Y | 6
  Epithelial microcystic edema indicator left eye: Baseline N, Post-Baseline Missing | 1
  Epithelial microcystic edema indicator left eye: Baseline Y, Post-Baseline N | 0
  Epithelial microcystic edema indicator left eye: Baseline Y, Post-Baseline Y | 0
  Epithelial microcystic edema indicator left eye: Baseline Y, Post-Baseline Missing | 0
  Epithelial microcystic edema indicator left eye: Baseline Missing, Post-Baseline N | 2
  Epithelial microcystic edema indicator left eye: Baseline Missing, Post-Baseline Y | 1
  Epithelial microcystic edema indicator left eye: Baseline Missing, Post-Baseline Missing | 1
  Epithelial microcystic edema indicator right eye: Baseline N, Post-Baseline N | 16
  Epithelial microcystic edema indicator right eye: Baseline N, Post-Baseline Y | 5
  Epithelial microcystic edema indicator right eye: Baseline N, Post-Baseline Missing | 1
  Epithelial microcystic edema indicator right eye: Baseline Y, Post-Baseline N | 0
  Epithelial microcystic edema indicator right eye: Baseline Y, Post-Baseline Y | 0
  Epithelial microcystic edema indicator right eye: Baseline Y, Post-Baseline Missing | 0
  Epithelial microcystic edema indicator right eye: Baseline Missing, Post-Baseline N | 3
  Epithelial microcystic edema indicator right eye: Baseline Missing, Post-Baseline Y | 2
  Epithelial microcystic edema indicator right eye: Baseline Missing, Post-Baseline Missing | 1
  Epithelial microcystic edema indicator worst eye: Baseline N, Post-Baseline N | 17
  Epithelial microcystic edema indicator worst eye: Baseline N, Post-Baseline Y | 6
  Epithelial microcystic edema indicator worst eye: Baseline N, Post-Baseline Missing | 1
  Epithelial microcystic edema indicator worst eye: Baseline Y, Post-Baseline N | 0
  Epithelial microcystic edema indicator worst eye: Baseline Y, Post-Baseline Y | 0
  Epithelial microcystic edema indicator worst eye: Baseline Y, Post-Baseline Missing | 0
  Epithelial microcystic edema indicator worst eye: Baseline Missing, Post-Baseline N | 2
  Epithelial microcystic edema indicator worst eye: Baseline Missing, Post-Baseline Y | 1
  Epithelial microcystic edema indicator worst eye: Baseline Missing, Post-Baseline Missing | 1
  Microcysts without edema indicator left eye: Baseline N, Post-Baseline N | 8
  Microcysts without edema indicator left eye: Baseline N, Post-Baseline Y | 15
  Microcysts without edema indicator left eye: Baseline N, Post-Baseline Missing | 1
  Microcysts without edema indicator left eye: Baseline Y, Post-Baseline N | 0
  Microcysts without edema indicator left eye: Baseline Y, Post-Baseline Y | 0
  Microcysts without edema indicator left eye: Baseline Y, Post-Baseline Missing | 0
  Microcysts without edema indicator left eye: Baseline Missing, Post-Baseline N | 0
  Microcysts without edema indicator left eye: Baseline Missing, Post-Baseline Y | 3
  Microcysts without edema indicator left eye: Baseline Missing, Post-Baseline Missing | 1
  Microcysts without edema indicator right eye: Baseline N, Post-Baseline N | 7
  Microcysts without edema indicator right eye: Baseline N, Post-Baseline Y | 14
  Microcysts without edema indicator right eye: Baseline N, Post-Baseline Missing | 1
  Microcysts without edema indicator right eye: Baseline Y, Post-Baseline N | 0
  Microcysts without edema indicator right eye: Baseline Y, Post-Baseline Y | 0
  Microcysts without edema indicator right eye: Baseline Y, Post-Baseline Missing | 0
  Microcysts without edema indicator right eye: Baseline Missing, Post-Baseline N | 1
  Microcysts without edema indicator right eye: Baseline Missing, Post-Baseline Y | 4
  Microcysts without edema indicator right eye: Baseline Missing, Post-Baseline Missing | 1
  Microcysts without edema indicator worst eye: Baseline N, Post-Baseline N | 8
  Microcysts without edema indicator worst eye: Baseline N, Post-Baseline Y | 15
  Microcysts without edema indicator worst eye: Baseline N, Post-Baseline Missing | 1
  Microcysts without edema indicator worst eye: Baseline Y, Post-Baseline N | 0
  Microcysts without edema indicator worst eye: Baseline Y, Post-Baseline Y | 0
  Microcysts without edema indicator worst eye: Baseline Y, Post-Baseline Missing | 0
  Microcysts without edema indicator worst eye: Baseline Missing, Post-Baseline N | 0
  Microcysts without edema indicator worst eye: Baseline Missing, Post-Baseline Y | 3
  Microcysts without edema indicator worst eye: Baseline Missing, Post-Baseline Missing | 1
  Corneal neovascularization indicator left eye: Baseline N, Post-Baseline N | 22
  Corneal neovascularization indicator left eye: Baseline N, Post-Baseline Y | 1
  Corneal neovascularization indicator left eye: Baseline N, Post-Baseline Missing | 2
  Corneal neovascularization indicator left eye: Baseline Y, Post-Baseline N | 0
  Corneal neovascularization indicator left eye: Baseline Y, Post-Baseline Y | 0
  Corneal neovascularization indicator left eye: Baseline Y, Post-Baseline Missing | 0
  Corneal neovascularization indicator left eye: Baseline Missing, Post-Baseline N | 2
  Corneal neovascularization indicator left eye: Baseline Missing, Post-Baseline Y | 1
  Corneal neovascularization indicator left eye: Baseline Missing, Post-Baseline Missing | 0
  Corneal neovascularization indicator right eye: Baseline N, Post-Baseline N | 20
  Corneal neovascularization indicator right eye: Baseline N, Post-Baseline Y | 1
  Corneal neovascularization indicator right eye: Baseline N, Post-Baseline Missing | 2
  Corneal neovascularization indicator right eye: Baseline Y, Post-Baseline N | 0
  Corneal neovascularization indicator right eye: Baseline Y, Post-Baseline Y | 1
  Corneal neovascularization indicator right eye: Baseline Y, Post-Baseline Missing | 0
  Corneal neovascularization indicator right eye: Baseline Missing, Post-Baseline N | 3
  Corneal neovascularization indicator right eye: Baseline Missing, Post-Baseline Y | 1
  Corneal neovascularization indicator right eye: Baseline Missing, Post-Baseline Missing | 0
  Corneal neovascularization indicator worst eye: Baseline N, Post-Baseline N | 21
  Corneal neovascularization indicator worst eye: Baseline N, Post-Baseline Y | 1
  Corneal neovascularization indicator worst eye: Baseline N, Post-Baseline Missing | 2
  Corneal neovascularization indicator worst eye: Baseline Y, Post-Baseline N | 0
  Corneal neovascularization indicator worst eye: Baseline Y, Post-Baseline Y | 1
  Corneal neovascularization indicator worst eye: Baseline Y, Post-Baseline Missing | 0
  Corneal neovascularization indicator worst eye: Baseline Missing, Post-Baseline N | 2
  Corneal neovascularization indicator worst eye: Baseline Missing, Post-Baseline Y | 1
  Corneal neovascularization indicator worst eye: Baseline Missing, Post-Baseline Missing | 0
  Subepithelial haze indicator left eye: Baseline N, Post-Baseline N | 16
  Subepithelial haze indicator left eye: Baseline N, Post-Baseline Y | 9
  Subepithelial haze indicator left eye: Baseline N, Post-Baseline Missing | 1
  Subepithelial haze indicator left eye: Baseline Y, Post-Baseline N | 1
  Subepithelial haze indicator left eye: Baseline Y, Post-Baseline Y | 0
  Subepithelial haze indicator left eye: Baseline Y, Post-Baseline Missing | 0
  Subepithelial haze indicator left eye: Baseline Missing, Post-Baseline N | 1
  Subepithelial haze indicator left eye: Baseline Missing, Post-Baseline Y | 0
  Subepithelial haze indicator left eye: Baseline Missing, Post-Baseline Missing | 0
  Subepithelial haze indicator right eye: Baseline N, Post-Baseline N | 16
  Subepithelial haze indicator right eye: Baseline N, Post-Baseline Y | 8
  Subepithelial haze indicator right eye: Baseline N, Post-Baseline Missing | 1
  Subepithelial haze indicator right eye: Baseline Y, Post-Baseline N | 1
  Subepithelial haze indicator right eye: Baseline Y, Post-Baseline Y | 0
  Subepithelial haze indicator right eye: Baseline Y, Post-Baseline Missing | 0
  Subepithelial haze indicator right eye: Baseline Missing, Post-Baseline N | 2
  Subepithelial haze indicator right eye: Baseline Missing, Post-Baseline Y | 0
  Subepithelial haze indicator right eye: Baseline Missing, Post-Baseline Missing | 0
  Subepithelial haze indicator worst eye: Baseline N, Post-Baseline N | 17
  Subepithelial haze indicator worst eye: Baseline N, Post-Baseline Y | 9
  Subepithelial haze indicator worst eye: Baseline N, Post-Baseline Missing | 1
  Subepithelial haze indicator worst eye: Baseline Y, Post-Baseline N | 0
  Subepithelial haze indicator worst eye: Baseline Y, Post-Baseline Y | 0
  Subepithelial haze indicator worst eye: Baseline Y, Post-Baseline Missing | 0
  Subepithelial haze indicator worst eye: Baseline Missing, Post-Baseline N | 1
  Subepithelial haze indicator worst eye: Baseline Missing, Post-Baseline Y | 0
  Subepithelial haze indicator worst eye: Baseline Missing, Post-Baseline Missing | 0

34. Secondary Outcome: Part 2 - Number of Participants With Worse Case Post-baseline Punctate Keratopathy Findings
Description: Participants with worse case punctate keratopathy findings post baseline at any ocular exam by right eye, left eye and worse eye are presented as none, mild, moderate and severe. Worse eye indicates the eye with the worst visual acuity. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 26
Participants
  Right eye, Worst findings: None | 2
  Right eye, Worst findings: Mild | 11
  Right eye, Worst findings: Moderate | 7
  Right eye, Worst findings: Severe | 6
  Left eye, Worst findings: None | 2
  Left eye, Worst findings: Mild | 9
  Left eye, Worst findings: Moderate | 9
  Left eye, Worst findings: Severe | 6
  Worst eye, Worst findings: None | 2
  Worst eye, Worst findings: Mild | 8
  Worst eye, Worst findings: Moderate | 10
  Worst eye, Worst findings: Severe | 6
  Right eye, Most frequent findings: None | 10
  Right eye, Most frequent findings: Mild | 14
  Right eye, Most frequent findings: Moderate | 2
  Right eye, Most frequent findings: Severe | 0
  Left eye, Most frequent findings: None | 8
  Left eye, Most frequent findings: Mild | 13
  Left eye, Most frequent findings: Moderate | 5
  Left eye, Most frequent findings: Severe | 0
  Worst eye, Most frequent findings: None | 7
  Worst eye, Most frequent findings: Mild | 14
  Worst eye, Most frequent findings: Moderate | 5
  Worst eye, Most frequent findings: Severe | 0

35. Secondary Outcome: Part 2 - Number of Participants With Worst-case Shift From Baseline in Lens Examinations
Description: Participants with worst-case shift from baseline in corneal examination which included: clear, pseudophakia, nuclear sclerosis, cortical cataract and posterior subcapsular cataract by right eye, left eye and worse eye are presented as yes (Y), no (N) and missing. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Participants
  Clear Indicator, Left eye: Baseline N, Post-Baseline N | 12
  Clear Indicator, Left eye: Baseline N, Post-Baseline Y | 0
  Clear Indicator, Left eye: Baseline N, Post-Baseline N=Missing | 3
  Clear Indicator, Left eye: Baseline Y, Post-Baseline N | 3
  Clear Indicator, Left eye: Baseline Y, Post-Baseline Y | 10
  Clear Indicator, Left eye: Baseline Y, Post-Baseline Missing | 0
  Clear Indicator, Left eye: Baseline Missing, Post-Baseline N | 0
  Clear Indicator, Left eye: Baseline Missing, Post-Baseline Y | 0
  Clear Indicator, Left eye: Baseline Missing, Post-Baseline Missing | 0
  Clear Indicator, Right eye: Baseline N, Post-Baseline N | 12
  Clear Indicator, Right eye: Baseline N, Post-Baseline Y | 0
  Clear Indicator, Right eye: Baseline N, Post-Baseline N=Missing | 3
  Clear Indicator, Right eye: Baseline Y, Post-Baseline N | 3
  Clear Indicator, Right eye: Baseline Y, Post-Baseline Y | 10
  Clear Indicator, Right eye: Baseline Y, Post-Baseline Missing | 0
  Clear Indicator, Right eye: Baseline Missing, Post-Baseline N | 0
  Clear Indicator, Right eye: Baseline Missing, Post-Baseline Y | 0
  Clear Indicator, Right eye: Baseline Missing, Post-Baseline Missing | 0
  Clear Indicator, worse eye: Baseline N, Post-Baseline N | 12
  Clear Indicator, worse eye: Baseline N, Post-Baseline Y | 0
  Clear Indicator, worse eye: Baseline N, Post-Baseline N=Missing | 3
  Clear Indicator, worse eye: Baseline Y, Post-Baseline N | 3
  Clear Indicator, worse eye: Baseline Y, Post-Baseline Y | 10
  Clear Indicator, worse eye: Baseline Y, Post-Baseline Missing | 0
  Clear Indicator, worse eye: Baseline Missing, Post-Baseline N | 0
  Clear Indicator, worse eye: Baseline Missing, Post-Baseline Y | 0
  Clear Indicator, worse eye: Baseline Missing, Post-Baseline Missing | 0
  Cortical Cataract Indicator, Left eye: Baseline N, Post-Baseline N | 7
  Cortical Cataract Indicator, Left eye: Baseline N, Post-Baseline Y | 3
  Cortical Cataract Indicator, Left eye: Baseline N, Post-Baseline N=Missing | 2
  Cortical Cataract Indicator, Left eye: Baseline Y, Post-Baseline N | 0
  Cortical Cataract Indicator, Left eye: Baseline Y, Post-Baseline Y | 2
  Cortical Cataract Indicator, Left eye: Baseline Y, Post-Baseline Missing | 1
  Cortical Cataract Indicator, Left eye: Baseline Missing, Post-Baseline N | 2
  Cortical Cataract Indicator, Left eye: Baseline Missing, Post-Baseline Y | 1
  Cortical Cataract Indicator, Left eye: Baseline Missing, Post-Baseline Missing | 10
  Cortical Cataract Indicator, Right eye: Baseline N, Post-Baseline N | 7
  Cortical Cataract Indicator, Right eye: Baseline N, Post-Baseline Y | 3
  Cortical Cataract Indicator, Right eye: Baseline N, Post-Baseline N=Missing | 1
  Cortical Cataract Indicator, Right eye: Baseline Y, Post-Baseline N | 0
  Cortical Cataract Indicator, Right eye: Baseline Y, Post-Baseline Y | 2
  Cortical Cataract Indicator, Right eye: Baseline Y, Post-Baseline Missing | 2
  Cortical Cataract Indicator, Right eye: Baseline Missing, Post-Baseline N | 3
  Cortical Cataract Indicator, Right eye: Baseline Missing, Post-Baseline Y | 0
  Cortical Cataract Indicator, Right eye: Baseline Missing, Post-Baseline Missing | 10
  Cortical Cataract Indicator, Worse eye: Baseline N, Post-Baseline N | 7
  Cortical Cataract Indicator, Worse eye: Baseline N, Post-Baseline Y | 3
  Cortical Cataract Indicator, Worse eye: Baseline N, Post-Baseline N=Missing | 2
  Cortical Cataract Indicator, Worse eye: Baseline Y, Post-Baseline N | 0
  Cortical Cataract Indicator, Worse eye: Baseline Y, Post-Baseline Y | 2
  Cortical Cataract Indicator, Worse eye: Baseline Y, Post-Baseline Missing | 1
  Cortical Cataract Indicator, Worse eye: Baseline Missing, Post-Baseline N | 2
  Cortical Cataract Indicator, Worse eye: Baseline Missing, Post-Baseline Y | 1
  Cortical Cataract Indicator, Worse eye: Baseline Missing, Post-Baseline Missing | 10
  Nuclear Sclerosis, Left eye: Baseline N, Post-Baseline N | 2
  Nuclear Sclerosis, Left eye: Baseline N, Post-Baseline Y | 1
  Nuclear Sclerosis, Left eye: Baseline N, Post-Baseline N=Missing | 0
  Nuclear Sclerosis, Left eye: Baseline Y, Post-Baseline N | 1
  Nuclear Sclerosis, Left eye: Baseline Y, Post-Baseline Y | 8
  Nuclear Sclerosis, Left eye: Baseline Y, Post-Baseline Missing | 3
  Nuclear Sclerosis, Left eye: Baseline Missing, Post-Baseline N | 2
  Nuclear Sclerosis, Left eye: Baseline Missing, Post-Baseline Y | 1
  Nuclear Sclerosis, Left eye: Baseline Missing, Post-Baseline Missing | 10
  Nuclear Sclerosis, Right eye: Baseline N, Post-Baseline N | 2
  Nuclear Sclerosis, Right eye: Baseline N, Post-Baseline Y | 1
  Nuclear Sclerosis, Right eye: Baseline N, Post-Baseline N=Missing | 0
  Nuclear Sclerosis, Right eye: Baseline Y, Post-Baseline N | 1
  Nuclear Sclerosis, Right eye: Baseline Y, Post-Baseline Y | 8
  Nuclear Sclerosis, Right eye: Baseline Y, Post-Baseline Missing | 3
  Nuclear Sclerosis, Right eye: Baseline Missing, Post-Baseline N | 3
  Nuclear Sclerosis, Right eye: Baseline Missing, Post-Baseline Y | 0
  Nuclear Sclerosis, Right eye: Baseline Missing, Post-Baseline Missing | 10
  Nuclear Sclerosis, Worse eye: Baseline N, Post-Baseline N | 2
  Nuclear Sclerosis, Worse eye: Baseline N, Post-Baseline Y | 1
  Nuclear Sclerosis, Worse eye: Baseline N, Post-Baseline N=Missing | 0
  Nuclear Sclerosis, Worse eye: Baseline Y, Post-Baseline N | 1
  Nuclear Sclerosis, Worse eye: Baseline Y, Post-Baseline Y | 8
  Nuclear Sclerosis, Worse eye: Baseline Y, Post-Baseline Missing | 3
  Nuclear Sclerosis, Worse eye: Baseline Missing, Post-Baseline N | 2
  Nuclear Sclerosis, Worse eye: Baseline Missing, Post-Baseline Y | 1
  Nuclear Sclerosis, Worse eye: Baseline Missing, Post-Baseline Missing | 10
  Posterior Subcapsular Cataract, Left eye: Baseline N, Post-Baseline N | 7
  Posterior Subcapsular Cataract, Left eye: Baseline N, Post-Baseline Y | 3
  Posterior Subcapsular Cataract, Left eye: Baseline N, Post-Baseline N=Missing | 0
  Posterior Subcapsular Cataract, Left eye: Baseline Y, Post-Baseline N | 0
  Posterior Subcapsular Cataract, Left eye: Baseline Y, Post-Baseline Y | 2
  Posterior Subcapsular Cataract, Left eye: Baseline Y, Post-Baseline Missing | 3
  Posterior Subcapsular Cataract, Left eye: Baseline Missing, Post-Baseline N | 1
  Posterior Subcapsular Cataract, Left eye: Baseline Missing, Post-Baseline Y | 2
  Posterior Subcapsular Cataract, Left eye: Baseline Missing, Post-Baseline Missing | 10
  Posterior Subcapsular Cataract, Right eye: Baseline N, Post-Baseline N | 7
  Posterior Subcapsular Cataract, Right eye: Baseline N, Post-Baseline Y | 1
  Posterior Subcapsular Cataract, Right eye: Baseline N, Post-Baseline N=Missing | 0
  Posterior Subcapsular Cataract, Right eye: Baseline Y, Post-Baseline N | 0
  Posterior Subcapsular Cataract, Right eye: Baseline Y, Post-Baseline Y | 4
  Posterior Subcapsular Cataract, Right eye: Baseline Y, Post-Baseline Missing | 3
  Posterior Subcapsular Cataract, Right eye: Baseline Missing, Post-Baseline N | 1
  Posterior Subcapsular Cataract, Right eye: Baseline Missing, Post-Baseline Y | 2
  Posterior Subcapsular Cataract, Right eye: Baseline Missing, Post-Baseline Missing | 10
  Posterior Subcapsular Cataract, Worse eye: Baseline N, Post-Baseline N | 6
  Posterior Subcapsular Cataract, Worse eye: Baseline N, Post-Baseline Y | 3
  Posterior Subcapsular Cataract, Worse eye: Baseline N, Post-Baseline N=Missing | 0
  Posterior Subcapsular Cataract, Worse eye: Baseline Y, Post-Baseline N | 0
  Posterior Subcapsular Cataract, Worse eye: Baseline Y, Post-Baseline Y | 4
  Posterior Subcapsular Cataract, Worse eye: Baseline Y, Post-Baseline Missing | 3
  Posterior Subcapsular Cataract, Worse eye: Baseline Missing, Post-Baseline N | 1
  Posterior Subcapsular Cataract, Worse eye: Baseline Missing, Post-Baseline Y | 1
  Posterior Subcapsular Cataract, Worse eye: Baseline Missing, Post-Baseline Missing | 10
  Pseudophakia, Left eye: Baseline N, Post-Baseline N | 11
  Pseudophakia, Left eye: Baseline N, Post-Baseline Y | 3
  Pseudophakia, Left eye: Baseline N, Post-Baseline N=Missing | 3
  Pseudophakia, Left eye: Baseline Y, Post-Baseline N | 1
  Pseudophakia, Left eye: Baseline Y, Post-Baseline Y | 10
  Pseudophakia, Left eye: Baseline Y, Post-Baseline Missing | 0
  Pseudophakia, Left eye: Baseline Missing, Post-Baseline N | 0
  Pseudophakia, Left eye: Baseline Missing, Post-Baseline Y | 0
  Pseudophakia, Left eye: Baseline Missing, Post-Baseline Missing | 0
  Pseudophakia, Right eye: Baseline N, Post-Baseline N | 12
  Pseudophakia, Right eye: Baseline N, Post-Baseline Y | 2
  Pseudophakia, Right eye: Baseline N, Post-Baseline N=Missing | 3
  Pseudophakia, Right eye: Baseline Y, Post-Baseline N | 1
  Pseudophakia, Right eye: Baseline Y, Post-Baseline Y | 10
  Pseudophakia, Right eye: Baseline Y, Post-Baseline Missing | 0
  Pseudophakia, Right eye: Baseline Missing, Post-Baseline N | 0
  Pseudophakia, Right eye: Baseline Missing, Post-Baseline Y | 0
  Pseudophakia, Right eye: Baseline Missing, Post-Baseline Missing | 0
  Pseudophakia, Worse eye: Baseline N, Post-Baseline N | 11
  Pseudophakia, Worse eye: Baseline N, Post-Baseline Y | 4
  Pseudophakia, Worse eye: Baseline N, Post-Baseline N=Missing | 3
  Pseudophakia, Worse eye: Baseline Y, Post-Baseline N | 0
  Pseudophakia, Worse eye: Baseline Y, Post-Baseline Y | 10
  Pseudophakia, Worse eye: Baseline Y, Post-Baseline Missing | 0
  Pseudophakia, Worse eye: Baseline Missing, Post-Baseline N | 0
  Pseudophakia, Worse eye: Baseline Missing, Post-Baseline Y | 0
  Pseudophakia, Worse eye: Baseline Missing, Post-Baseline Missing | 0

36. Secondary Outcome: Part 2 - Percentage of Participants With Clinical Benefit Rate
Description: Clinical benefit rate was defined as the percentage of participants with a confirmed minimal response (MR) or better according to the IMWG Response Criteria. MR is >= 25% but < 49% reduction of serum M-protein and reduction in 24-hour urinary M-protein by 50-89%.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Percentage of Participants | 43 [24.5 to 62.8]

37. Secondary Outcome: Part 2 - Duration of Response
Description: Duration of response was defined as the time from first documented evidence of PR or better, to the time when disease progression (PD) is documented per IMWG response criteria; or death due to PD occurs among participants who achieve an overall response, i.e. confirmed PR or better. PD= Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 g/dL; Serum M-protein increase >= 1 g/dL if the lowest M-component was >=5 g/dL; Urinary M-protein (absolute increase must be >= 200 mg per 24 h). PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥ 90% or to <200 mg/24 h.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 12
Months | 7.6 [1.4 to NA] — The upper limit of 95% CI was not estimate due to limited number of events

38. Secondary Outcome: Part 2 - Time to Response
Description: Time to response (TTR) was defined as the time between the date of first dose and the first documented evidence of response (PR or better) among participants who achieved a confirmed response of PR or better.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 12
Months | 0.7 [0.7 to 1.4]

39. Secondary Outcome: Part 2 - Time to Best Response
Description: Time to best response was defined as the time between the date of first dose and the first best documented response (PR or better) among participants who achieved a confirmed response of PR or better.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Months
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 12
Months | 1.7 [0.7 to 5.6]

40. Secondary Outcome: Part 2 - Progression-free Survival
Description: Progression-free survival was defined as the time from first dose until the earliest date of PD per IMWG response criteria, or death due to any cause. PD= Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 g/dL; Serum M-protein increase >= 1 g/dL if the lowest M-component was >=5 g/dL; Urinary M-protein (absolute increase must be >= 200 mg per 24 h).
Time Frame: Up to approximately 178 weeks
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Months | 2.5 [0.8 to 5.6]

41. Secondary Outcome: Part 2 - Time to Disease Progression
Description: Time to disease progression was defined as the time from first dose until the earliest date of PD per IMWG response criteria, or death due to PD. PD= Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 g/dL; Serum M-protein increase >= 1 g/dL if the lowest M-component was >=5 g/dL; Urinary M-protein (absolute increase must be >= 200 mg per 24 h).
Time Frame: Up to approximately 178 weeks
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Months | 2.5 [0.8 to 5.6]

42. Secondary Outcome: Part 2 - Overall Survival
Description: Overall Survival was defined as the time from first dose until death due to any cause.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Months | NA [19.1 to NA] — The median and upper limit of 95% CI was not estimate due to limited number of events

43. Secondary Outcome: Part 1 - Maximum Concentration (Cmax) for Belantamab Mafodotin After First Dose
Description: Blood samples were collected for Pharmacokinetic (PK) analysis of belantamab mafodotin when administered intravenously in combination with pembrolizumab. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, end of infusion (EOI), 2, 4, 9, and 24 h post-SOI (start of infusion) on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: Pharmacokinetic (PK) Population included participants in the all treated population from whom at least one PK sample was obtained and analyzed for belantamab mafodotin. Due to bioanalytical issues, PK data were not collected and analyzed for belantamab mafodotin. Therefore, this PK parameter was not reported in this study.
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: Part 2 - Cmax for Belantamab Mafodotin After First Dose
Description: Blood samples were collected for PK analysis of belantamab mafodotin when administered intravenously in combination with pembrolizumab. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: Pharmacokinetic Population. Due to bioanalytical issues, PK data were not collected and analyzed for belantamab mafodotin. Therefore, this PK parameter was not reported in this study
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 0

45. Secondary Outcome: Part 1 - End of Infusion Concentration (C-EOI) for Belantamab Mafodotin
Description: as for outcome 44
Time Frame: EOI post belantamab mafodotin dose on Day 1 of each 21 day Cycle till Cycle 11
Population: as for outcome 44
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 0 | 0

46. Secondary Outcome: Part 2 - C-EOI for Belantamab Mafodotin
Description: as for outcome 44
Time Frame: EOI post belantamab mafodotin dose on Day 1 of each 21 day Cycle till Cycle 11
Population: as for outcome 44
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 0

47. Secondary Outcome: Part 1 - Time of Cmax (Tmax) for Belantamab Mafodotin After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: as for outcome 44
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 0 | 0

48. Secondary Outcome: Part 2 - Tmax for Belantamab Mafodotin After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: as for outcome 44
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 0

49. Secondary Outcome: Part 1 - Trough Concentration Prior to the Next Dose for Each Cycle (Ctrough) for Belantamab Mafodotin
Description: Blood samples were collected for PK analysis of belantamab mafodotin when administered intravenously in combination with pembrolizumab. Ctrough was calculated as the observed concentration at the end of a dosing interval, immediately before next study drug administration on Day 1 of each Cycle. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose on Day 1 of each 21 day cycle from Cycle 1 until Cycle 13
Population: as for outcome 44
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 0 | 0

50. Secondary Outcome: Part 2 - Ctrough for Belantamab Mafodotin
Description: as for outcome 49
Time Frame: Pre-dose on Day 1 of each 21 day cycle from Cycle 1 until Cycle 13
Population: as for outcome 44
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 0

51. Secondary Outcome: Part 1 - Last Time Point Where the Concentration is Above the Limit of Quantification (Tlast) for Belantamab Mafodotin After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: as for outcome 44
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 0 | 0

52. Secondary Outcome: Part 2 - Tlast for Belantamab Mafodotin After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: as for outcome 44
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 0

53. Secondary Outcome: Part 1 - Area Under Plasma Concentration-time Curve (AUC) From Time 0 to End of the Dosing Interval [AUC (0-tau)] for Belantamab Mafodotin After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: as for outcome 44
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 0 | 0

54. Secondary Outcome: Part 2 - AUC (0-tau) for Belantamab Mafodotin After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: as for outcome 44
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 0

55. Secondary Outcome: Part 1 - Cmax for Total Monoclonal Antibody (mAb) After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 hour post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 4 | 7
ug/mL | 43.57 (7.1) | 64.45 (21.5)

56. Secondary Outcome: Part 2 - Cmax for Total mAb After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, and 24 hour post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 26
ug/mL | 46.70 (23.3)

57. Secondary Outcome: Part 1 - C-EOI for Total mAb
Description: as for outcome 44
Time Frame: EOI post belantamab mafodotin dose on Day 1 of Cycle 1, Cycle 2, Cycle 5, Cycle 8, and Cycle 11
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 4 | 7
ug/mL
  Cycle 1 | 40.15 [36.3 to 44.4] | 65.30 [44.6 to 73.5]
  Cycle 2: number analyzed (Participants) | 4 | 4
  Cycle 2 | 53.90 [39.1 to 66.3] | 64.65 [16.1 to 90.1]
  Cycle 5: number analyzed (Participants) | 4 | 3
  Cycle 5 | 54.65 [46.5 to 78.2] | 73.90 [42.6 to 101.0]
  Cycle 8: number analyzed (Participants) | 1 | 2
  Cycle 8 | 63.70 [63.70 to 63.70] | 39.75 [12.9 to 66.6]
  Cycle 11: number analyzed (Participants) | 1 | 1
  Cycle 11 | 65.40 [65.40 to 65.40] | 54.80 [54.80 to 54.80]

58. Secondary Outcome: Part 2 - C-EOI for Total mAb
Description: as for outcome 44
Time Frame: EOI post belantamab mafodotin dose on Day 1 of Cycle 1, Cycle 2, and Cycle 5
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 23
ug/mL
  Cycle 1: number analyzed (Participants) | 21
  Cycle 1 | 48.60 [17.4 to 68.9]
  Cycle 2 | 53.00 [26.5 to 71.1]
  Cycle 5: number analyzed (Participants) | 6
  Cycle 5 | 52.35 [36.9 to 70.5]

59. Secondary Outcome: Part 1 - Tmax for Total mAb After First Dose
Description: as for outcome 44
Time Frame: as for outcome 55
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 4 | 7
Hour | 1.100 [0.53 to 2.18] | 1.520 [0.75 to 2.05]

60. Secondary Outcome: Part 2 - Tmax for Total mAb After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, and 24 hour post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 26
Hour | 0.945 [0.47 to 2.33]

61. Secondary Outcome: Part 1 - Ctrough for Total mAb
Description: as for outcome 49
Time Frame: Cycle 1, Cycle 4, Cycle 7, Cycle 10, and Cycle 13
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 5 | 4
ug/mL
  Cycle 1: number analyzed (Participants) | 3 | 4
  Cycle 1 | 5.420 [3.85 to 7.87] | 13.350 [1.83 to 13.50]
  Cycle 4: number analyzed (Participants) | 5 | 2
  Cycle 4 | 8.91 [0 to 30.8] | 18.80 [18.1 to 19.5]
  Cycle 7: number analyzed (Participants) | 1 | 2
  Cycle 7 | 26.90 [26.9 to 26.9] | 45.05 [23.9 to 66.2]
  Cycle 10: number analyzed (Participants) | 1 | 1
  Cycle 10 | 18.40 [18.4 to 18.4] | 21.70 [21.7 to 21.7]
  Cycle 13: number analyzed (Participants) | 2 | 0
  Cycle 13 | 18.05 [18.0 to 18.1] |

62. Secondary Outcome: Part 2 - Ctrough for Total mAb
Description: as for outcome 49
Time Frame: Cycle 1 and Cycle 4
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 20
ug/mL
  Cycle 1 | 7.735 [1.28 to 12.70]
  Cycle 4: number analyzed (Participants) | 7
  Cycle 4 | 11.60 [9.15 to 31.0]

63. Secondary Outcome: Part 1 - Last Time Point Where the Concentration is Above the Limit of Quantification (Tlast) for Total mAb After First Dose
Description: Blood samples were collected for PK analysis of belantamab mafodotin when administered intravenously in combination with pembrolizumab. PK parameter was determined using standard non-compartmental methods. Tlast is the time of last observed quantifiable concentration of belantamab mafodotin in Cycle 1 which extended beyond protocol defined duration for some participants across treatment groups.
Time Frame: as for outcome 55
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 5 | 7
Hour | 501.800 [70.03 to 507.23] | 481.580 [72.27 to 551.80]

64. Secondary Outcome: Part 2 - Tlast for Total mAb After First Dose
Description: as for outcome 63
Time Frame: Pre-dose, EOI, 2, 4, and 24 hour post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Hour | 503.140 [72.50 to 2060.68]

65. Secondary Outcome: Part 1 - AUC (0-tau) for Total mAb After First Dose
Description: as for outcome 44
Time Frame: as for outcome 55
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 3 | 4
h*ug/mL | 6237.2 (17.9) | 10817.8 (48.5)

66. Secondary Outcome: Part 2 - AUC (0-tau) for Total mAb After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, and 24 hour post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 19
h*ug/mL | 7949.0 (27.2)

67. Secondary Outcome: Part 1 - Cmax for Cysteine Maleimidocaproyl Monomethyl Auristatin F (Cys-mcMMAF) After First Dose
Description: as for outcome 44
Time Frame: as for outcome 55
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 2 | 5
ng/mL | 1.5799 (30.4) | 1.0966 (40.9)

68. Secondary Outcome: Part 2 - Cmax for Cys-mcMMAF After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, and 24 hour post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 26
ng/mL | 1.2481 (111.5)

69. Secondary Outcome: Part 1 - C-EOI for Cys-mcMMAF After First Dose
Description: as for outcome 44
Time Frame: EOI post belantamab mafodotin dose on Day 1 of Cycle 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 2 | 7
ng/mL | 0.7110 [0.342 to 1.080] | 0.7630 [0.169 to 1.980]

70. Secondary Outcome: Part 2 - C-EOI for Cys-mcMMAF After First Dose
Description: as for outcome 44
Time Frame: EOI post belantamab mafodotin dose on Day 1 of Cycle 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 25
ng/mL | 0.3150 [0.131 to 20.300]

71. Secondary Outcome: Part 1 - Tmax for Cys-mcMMAF After First Dose
Description: as for outcome 63
Time Frame: as for outcome 55
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 2 | 5
Hour | 13.510 [4.05 to 22.97] | 4.120 [0.57 to 73.03]

72. Secondary Outcome: Part 2 - Tmax for Cys-mcMMAF After First Dose
Description: as for outcome 63
Time Frame: Pre-dose, EOI, 2, 4, and 24 hour post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 26
Hour | 23.580 [0.52 to 70.65]

73. Secondary Outcome: Part 1 - Tlast for Cys-mcMMAF After First Dose
Description: as for outcome 63
Time Frame: as for outcome 55
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 3 | 7
Hour | 161.380 [70.03 to 168.13] | 171.250 [72.27 to 501.28]

74. Secondary Outcome: Part 2 - Tlast for Cys-mcMMAF After First Dose
Description: as for outcome 63
Time Frame: Pre-dose, EOI, 2, 4, and 24 hour post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hour
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 28
Hour | 167.510 [23.90 to 503.15]

75. Secondary Outcome: Part 1 - AUC From Time 0 to 168 h After Dosing [AUC (0-168h)] for Cys-mcMMAF After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 hour post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, and Cycle 1 Day 8
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 1 | 4
h*ug/mL | 155.27 | 90.61 (34.5)

76. Secondary Outcome: Part 2 - AUC (0-168 h) for Cys-mcMMAF After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, and 24 hour post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, and Cycle 1 Day 8
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 18
h*ug/mL | 128.38 (70.9)

77. Secondary Outcome: Part 1 - Cmax for Pembrolizumab After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: Pharmacokinetic Population. Pembrolizumab data were not collected and analyzed. Therefore, this PK parameter was not reported in this study.
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 0 | 0

78. Secondary Outcome: Part 2 - Cmax for Pembrolizumab After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: as for outcome 77
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 0

79. Secondary Outcome: Part 1 - Tmax for Pembrolizumab After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: as for outcome 77
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 0 | 0

80. Secondary Outcome: Part 2 - Tmax for Pembrolizumab After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: as for outcome 77
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 0

81. Secondary Outcome: Part 1 - AUC (0-tau) for Pembrolizumab After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: as for outcome 77
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 0 | 0

82. Secondary Outcome: Part 2 - AUC (0-tau) for Pembrolizumab After First Dose
Description: as for outcome 44
Time Frame: Pre-dose, EOI, 2, 4, 9, and 24 h post-SOI on Cycle 1 Day 1, Cycle 1 Day 4, Cycle 1 Day 8, and pre-dose on Cycle 2 Day 1
Population: as for outcome 77
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 0

83. Secondary Outcome: Part 1 - Number of Participants With Post-baseline Positive Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples collected for the analysis of the presence of ADAs using validated immunoassays. All samples were tested in screening assay, and positive samples were further characterized for antibody titers. At the time of primary results posting, there was no participants with positive ADA results. Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Baseline (Day 1) and until end of treatment (up to 178 weeks)
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 4 | 7
Participants
  Baseline | 0 | 0
  End of Treatment: number analyzed (Participants) | 4 | 5
  End of Treatment | 0 | 0

84. Secondary Outcome: Part 2 - Number of Participants With Post-baseline Positive ADAs Against Belantamab Mafodotin
Description: as for outcome 83
Time Frame: Baseline (Day 1) and until end of treatment (up to 178 weeks)
Population: All Treated Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 27
Participants
  Baseline | 0
  End of Treatment: number analyzed (Participants) | 18
  End of Treatment | 0

85. Secondary Outcome: Part 1 - Titers of ADAs Against Belantamab Mafodotin
Description: Serum samples collected for the analysis of the presence of ADAs using validated immunoassays. All samples were to be further tested in screening assay, and positive samples were further to be characterized for antibody titers.
Time Frame: Up to approximately 178 weeks
Population: All Treated Population. There were no participants with positive ADA results. Hence the titer (concentration) of ADA was not collected.
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation
Number analyzed (Participants) | 0 | 0

86. Secondary Outcome: Part 2 - Titers of ADAs Against Belantamab Mafodotin
Description: as for outcome 85
Time Frame: Baseline (Day 1) and up to approximately 178 weeks
Population: as for outcome 85
Arm/Group | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected from day 1 to week 178 for Main Study Phase and from week 178 to week 221 for PACT phase.
Description: All Treated Population included all participants who received at least one dose of study treatment.
Arm/Group | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion | PACT Phase- Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 2/6 | 3/7 | 7/28 | 0/2
Serious Adverse Events (participants affected / at risk) | 4/6 | 5/7 | 5/28 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 6/7 | 27/28 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation (N=6) | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation (N=7) | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion (N=28) | PACT Phase- Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Leishmaniasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (2) | 4 (6) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study Phase- Part 1: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Escalation (N=6) | Main Study Phase- Part 1: Belantamab Mafodotin 3.4 mg/kg + Pembrolizumab 200 mg Escalation (N=7) | Main Study Phase- Part 2: Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg Expansion (N=28) | PACT Phase- Belantamab Mafodotin 2.5 mg/kg + Pembrolizumab 200 mg (N=2)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 3 (3) | 5 (5) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 2 (4) | 2 (5) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 3 (6) | 9 (10) | 0 (0)
Blepharitis (Eye disorders) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 3 (4) | 1 (2) | 4 (4) | 0 (0)
Eye pruritus (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Keratopathy (Eye disorders) | 6 (7) | 6 (7) | 20 (27) | 0 (0)
Photophobia (Eye disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Vision blurred (Eye disorders) | 3 (4) | 2 (2) | 10 (10) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (2) | 7 (7) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Fatigue (General disorders) | 3 (9) | 3 (5) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 10 (12) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 7 (7) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Visual acuity tests abnormal (Investigations) | 1 (2) | 1 (2) | 1 (5) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (4) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT03848845/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT03848845/SAP_001.pdf